CLINICAL TRIAL: NCT03014999
Title: Corticospinal Excitability After rTMS in Spinal Cord Injury Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, PhD, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CNSexcit_SCI
Record Dates: First submitted 2016-10-02; First posted 2017-01-09 (Estimated); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Spinal Cord Injury
Keywords: Transcranial Magnetic Stimulation; Spinal Cord Injury; Humans
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High frequency rTMS (Experimental): Volunteers will be submitted to high frequency of repetitive transcranial magnetic stimulation (10Hz)
  Interventions: Device: High frequency rTMS (repetitive Transcranial Magnetic Stimulation)
- Low frequency rTMS (Experimental): Volunteers will be submitted to low frequency of repetitive transcranial magnetic stimulation (1Hz)
  Interventions: Device: Low frequency rTMS (repetitive Transcranial Magnetic Stimulation)
- Sham rTMS (Sham Comparator): Volunteers will be submitted to sham session of repetitive transcranial magnetic stimulation
  Interventions: Device: sham rTMS (repetitive Transcranial Magnetic Stimulation)

INTERVENTIONS:
Device: High frequency rTMS (repetitive Transcranial Magnetic Stimulation) — Higher cortical representation area of first right dorsal interosseous muscle will be determined through a figure-eight coil connected to the magnetic stimulator (Rapid2, Magstim, UK) held manually and at 45 degrees from the midline over the right primary motor cortex (C3 - 10/20 System). Then, will be determined the rest motor threshold by finding the lowest stimulator output that elicit motor evoked potential at least 50μV. After determined the RMT, the coil will be positioned over the scalp (Cz - 10/20 System). Thereafter, RMT will be measure. rTMS protocols was based on previous studies. High frequency protocol: 10Hz, 90% RMT, 45 trains, 40 stimuli per train, inter interval of 28s, 1800 stimuli. After each rTMS session, presence of adverse effects will be computed.
  Other Names: High frequency rTMS
  Arms: High frequency rTMS
Device: Low frequency rTMS (repetitive Transcranial Magnetic Stimulation) — Initially, the higher cortical representation area (hotspot) of first right dorsal interosseous (FDI) muscle will be determined through a figure-eight coil connected to the magnetic stimulator (Rapid2, Magstim, UK) held manually and at 45 degrees from the midline, will be placed over the right primary motor cortex (C3 - 10/20 System). Then, will be determined the rest motor threshold (RMT) by finding the lowest stimulator output that elicit motor evoked potential (MEP) at least 50 microvolts (μV). After determined the RMT, the coil will be positioned over the scalp (Cz - 10/20 System). Thereafter, RMT will be measure. Low frequency protocol: 1Hz, 90% RMT, 1500 stimuli (1 train). After each rTMS session, presence of adverse effects will be computed
  Other Names: Low frequency rTMS
  Arms: Low frequency rTMS
Device: sham rTMS (repetitive Transcranial Magnetic Stimulation) — The hotspot of first right dorsal interosseous (FDI) muscle will be determinate through a figure-eight coil connected to the magnetic stimulator positioned over the motor primary cortex (C3). Then, the motor threshold (RMT) of FDI will be measure. Sham rTMS will be performed with low frequency (1Hz, 90% RMT, 1500 stimuli) protocol using two coils. The first one - connected to the stimulator - will be positioned on a coil support close to the volunteer but not visible. Therefore, characteristic stimulation noises will be audible. The second - disconnected to the stimulator - will be placed over primary motor area Cz. After each rTMS session, presence of adverse effects will be computed.
  Other Names: sham rTMS
  Arms: Sham rTMS

SUMMARY:
A crossover trial with spinal cord injury volunteers will be conducted. Three sessions will be performed once a week in a counterbalanced order and at least with seven days washout period to minimize carry-over effects. In each session, volunteers will be submitted to quantity and quality of sleep, type of eating, fatigue and motivation level, Ashworth scale spasticity, cortical brain activity measures through simple pulse transcranial magnetic stimulation (pTMS), spinal cord activity measures through electrical stimulation and non-invasive brain stimulation (rTMS)

DETAILED DESCRIPTION:
After given prior informed consent, volunteers will be submitted to three randomized and counterbalanced sessions using a website (randomization.com) by a non-involved researcher. At study beginning, volunteers will be evaluated through structured questionnaire and each session, will comprise the following experimental sequence:

1. Quantity and quality of sleep: It will be enquired how many hours the volunteer slept in the last night. The quality of the sleep will be measured through an analogue scale graded from 0 (worst quality of sleep) to 10 points (best quality of sleep).
2. Type of eating: All the individuals will be asked about ingestion of food and drinks that could change the cortical excitability (e. g.; coffee, chocolate, energetic, soda e etcc). If positive, researchers will record the time since of ingestion and quantify the amount of food.
3. Fatigue and motivation level: It will be measured through an analogue scale graded from 0 (lower fatigue or motivation levels) to 10 points (greater fatigue or motivation levels).
4. Spasticity: It will be assessed by the modified Ashworth scale ranging from 0 to 4. Performs the passive drive member to be measured and observing the time it arises the resistance difficult the passive movement. This scale will be tested bilaterally in the muscles of the lower limbs, the tested muscles are the quadriceps, adductors, hamstring, dorsiflexors, hip flexors and flexors plant. The scale always applies by the same evaluator.
5. Spinal cord activity: the level of excitability of spinal cord will be measured through the following outcomes:

   • Hoffman reflex (H reflex): the H reflex will be elicited by a percutaneous electrical stimulation on tibial nerve delivered on popliteal fossa and recorded the electromyographic responses from the soleus muscle. The values of maximal H reflex, M wave and maximal H reflex and maximal M wave ratio (H/M ratio) will be obtained through a recruitment curve.

   The recruitment curve will start with a stimulus intensity delivered from 2 milliampere (mA) and increasing on steps of 1 mA until to M wave curve stabilization (no increasing of the M wave amplitude).

   • Homosynaptic depression (HD): the HD will be obtained through a serie of two consecutive stimuli separated by a interstimulus interval (from 30 ms until 10.000 ms). The stimuli will be delivered on popliteal fossa and the electromyographic responses from soleus muscle will be recorded. The stimuli will be delivered with the intensity necessary to produce the maximal H reflex (this information will be available in the recruitment curve as stated before). The difference between the first and the second stimuli for each interstimulus interval will give rise to the recovery curve.
6. Cortical excitability: the cortical excitability will be measured through the motor evoked potential (MEP) through simple pulse transcranial magnetic stimulation (BiStim2, Magstim, UK) Initially, the higher cortical representation area (hotspot) of first right dorsal interosseous (FDI) muscle will be determined through a figure-eight coil connected to the magnetic stimulator held manually at 45 degrees from the midline, will be placed over the right primary motor cortex (C3 - 10/20 System). Then, will be determined the rest motor threshold (RMT) by finding the lowest stimulator output that elicit motor evoked potential (MEP) at least 50 microvolts (μV). After determined the RMT, the MEP value will be obtained through twenty suprathreshold (130% of RMT) stimuli that will be delivered on primary motor cortex (C3).
7. rTMS: Initially, the higher cortical representation area (hotspot) of first right dorsal interosseous (FDI) muscle will be determined through a figure-eight coil connected to the magnetic stimulator (Rapid2, Magstim, UK) held manually at 45 degrees from the midline, will be placed over the right primary motor cortex (C3 - 10/20 System). Then, will be determined the rest motor threshold (RMT) by finding the lowest stimulator output that elicit motor evoked potential (MEP) at least 50 microvolts (μV). After determined the RMT, the coil will be positioned over the scalp (Cz - 10/20 System) and based on previous studies will be performed rTMS protocols. Low frequency protocol: 1 hertz (Hz), 90% RMT, 1500 stimuli (1 train). High frequency protocol: 10 Hz, 90% RMT, 45 trains, 40 stimuli per train, inter interval of 28 seconds, 1800 stimuli. Sham rTMS will be performed with low frequency protocol using two coils. The first one - connected to the stimulator - will be positioned on a coil support close to the volunteer but not visible. Therefore, characteristic stimulation noises will be audible. The second - disconnected to the stimulator - will be placed over left primary motor area. After each rTMS session, presence of adverse effects will be computed.
8. Spasticity: this evaluation will be performed immediately after (T0), thirty minutes after (T1) and 1 hour after (T2) the rTMS. The procedures will be conducted following the same protocol.
9. Spinal cord activity: this evaluation will be performed immediately after (T0), thirty minutes after (T1) and 1 hour after (T2) the rTMS. The procedures will be conducted following the same protocol.
10. Cortical brain activity: this evaluation will be performed after each revaluation of spinal cord activity (T0, T1 and T2). The procedures will be conducted following the same protocol.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed (assessed by Edinburgh Handedness Inventory)
* Incomplete Spinal cord injury thoracic or lombar levels
* Sensorio-motor impairment C or D according to American Spinal Cord Injury Association (ASIA)
* To be on chronic stage of injury (> 8 months);
* Strength grade of hip flexors and knee extensors ≥ 1 according to Medical Research Council;
* Not to be a community walker

Exclusion Criteria:

* Pregnancy
* Presence of metallic implant close to the target stimulation area
* Acute eczema under the target stimulation area
* Pacemaker
* History of seizures or epilepsy
* Hemodynamic instability
* History of neurological or orthopedic disease not related to spinal cord injury
* Cognitive impairment
* knee, ankle or hip flexor contracture superior to 20º;
* Changes on medication during the study execution

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Spasticity | three weeks (during stimulation protocol)
  Assessment by modified ashworth scale
Spinal excitability | three weeks (during stimulation protocol)
  Spinal excitability measures will be assessed by electrical stimulation of the tibial nerve (H-reflex and homosynaptic depression). The volunteer should stay in prone position for the stimulation of the tibial nerve (in the region of the popliteal fossa). The spinal cord excitability will be assessed by Hoffman reflex (Hr) and homosynaptic depression (DH) before intervention and immediately, 30 and 60 minutes after. The ration of maximal Hr/ maximal M-wave amplitude and interestimulus interval of 150ms, 200ms, 250 ms and 300ms of the Hr recovery curve were observed when assessing outcome data.

SECONDARY OUTCOMES:
Cortical excitability | three weeks (during stimulation protocol)
  The motor evoked potential (MEP) will be provided by twenty unconditioned stimuli (130% RMT)

CONTACTS AND LOCATIONS:
Overall Officials: Kátia M Silva, PhD, Study Director — Universidade Federal de Pernambuco
Locations (1):
- Federal University of Pernambuco, Applied Neuroscience Laboratory, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No